CLINICAL TRIAL: NCT04675372
Title: Based on the Real-time Monitoring of Nociceptive Index, Dexmedetomidine as a Neuraxial Adjuvant Facilitate Analgesia
Brief Title: Dexmedetomidine Facilitate Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IRB-XWAD-202008-12
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Lower Limb Fracture; Nerve Block
Keywords: Dexmedetomidine; nociceptive index
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Dexmedetomidine group (Group DEX) was given 1.5ug/kg/h Dexmedetomidine continuous infusion Dexmedetomidine group (Group DEX)
  Interventions: Drug: Dexmedetomidine
- Group 2 (Active Comparator): Midazolam group (Group MID) was continuously pumped with 0.05mg/kg/h midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine group (Group D) was given 1.5ug/kg/h Dexmedetomidine continuous infusion
  Arms: Group 1
Drug: Midazolam — Midazolam group (Group M) was continuously pumped with 0.05mg/kg/h midazolam
  Arms: Group 2

SUMMARY:
Pre-clinic evidences showed that DEX produces antinociception by inhibiting the activation of spinal microglia and astrocyte decreasing noxious stimuli evoked release of nociceptive substances and further interrupting the spinal neuron-glia cross talk and regulating the nociceptive transmission under chronic pain condition. in this study, the analgesic efficacy of Dexmedetomidine was evaluated by a new non-invasive nociceptive index (qNOX). In this study, Anagel6000 analgesia monitor was used to quantitatively compare the analgesic efficacy of Dexmedetomidine compared with Midazolam.

DETAILED DESCRIPTION:
Pre-clinic evidences showed that DEX produces antinociception by inhibiting the activation of spinal microglia and astrocyte decreasing noxious stimuli evoked release of nociceptive substances and further interrupting the spinal neuron-glia cross talk and regulating the nociceptive transmission under chronic pain condition. in this study, the analgesic efficacy of Dexmedetomidine was evaluated by a new non-invasive nociceptive index (qNOX). In this study, Anagel6000 analgesia monitor was used to quantitatively compare the analgesic efficacy of Dexmedetomidine compared with Midazolam.

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 80 years old
* American Association of anesthesiologists (ASA) grade Ⅱ ~ IV
* body mass index (BMI) 18.5-40
* planning undergoing peripheral nerve block

Exclusion Criteria:

* incomplete effect of nerve block
* Alzheimer's disease
* implanted cardiac pacemakers
* mental illness
* epilepsy
* autonomic nervous system diseases
* projected the duration of the operation was more than 3 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
nociceptive index | During operation
  qNOX reached target 80 during drug infusion（qNOX<80 Adequate；qNOX>80 unadequate）

SECONDARY OUTCOMES:
hypoxemia | During operation
  incidence of hypoxemia(SPO2<95%Mild hypoxemia,SPO2<90% moderate hypoxemia, SPO2<85% severe hypoxemia)
systolic blood pressure | During operation
  Change of systolic blood pressure(SBP)
heart rate | During operation
  fluctuation of heart rate(HR)
diastolic blood pressure | During operation
  fluctuation of diastolic blood pressure(DBP)
muscular activity | During operation
  fluctuation of muscular activity (EMG)

CONTACTS AND LOCATIONS:
Locations (1):
- China International Neuroscience, Beijing, Beijing Municipality, China